CLINICAL TRIAL: NCT05631093
Title: A Phase 3, Randomized, Active-Controlled, Open-Label Clinical Study to Evaluate a Switch to Doravirine/Islatravir (DOR/ISL 100 mg/0.25 mg) Once-Daily in Participants With HIV-1 Who Are Virologically Suppressed on Antiretroviral Therapy
Brief Title: A Switch to Doravirine/Islatravir (DOR/ISL) in Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Who Are Virologically Suppressed on Antiretroviral Therapy (ART) (MK-8591A-051)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8591A-051; MK-8591A-051 (Other: MSD); jRCT2031220698 (Registry Identifier: jRCT); U1111-1283-3894 (Registry Identifier: UTN); 2022-502127-22-00 (Registry Identifier: EU CT); 2022-502127-22 (EudraCT Number)
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DOR/ISL (Experimental): Participants with Human Immunodeficiency Virus-1 (HIV-1) that have been virologically suppressed for ≥3 consecutive months who were previously treated with continuous baseline antiretroviral therapy (ART) receive doravine/islatravir (DOR/ISL), a fixed dose combination (FDC) of 100 mg DOR/0.25 mg ISL orally once daily (qd) for 144 weeks. At Week 144, participants who consent to enter the optional study extension will continue to receive DOR/ISL qd (100 mg/0.25 mg) for an additional 96 weeks or until it is commercially accessible (whichever comes first).
  Interventions: Drug: DOR/ISL
- ART + DOR/ISL (Active Comparator): Participants with HIV-1 that has been virologically suppressed for ≥3 consecutive months who were previously treated with continuous baseline ART received standard of care (SOC) ART for 48 weeks, followed by treatment with DOR/ISL as a FDC of 100 mg DOR/0.25 mg ISL orally qd until Week 144. At Week 144, participants who consent to enter the optional study extension will continue to receive DOR/ISL qd (100 mg/0.25 mg) for an additional 96 weeks or until it is commercially accessible (whichever comes first).
  Interventions: Drug: ART

INTERVENTIONS:
Drug: ART — Standard of care ART, per approved product list, taken orally
  Arms: ART + DOR/ISL
Drug: DOR/ISL — Single tablet combination of 100 mg doravirine (DOR) with 0.25 mg Islatravir (ISL) in tablet form, taken orally, once daily.
  Other Names: MK-8591A
  Arms: DOR/ISL

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of a switch to Doravirine/Islatravir (DOR/ISL) compared with continued baseline antiretroviral therapy (ART), through Week 48; and to evaluate the antiretroviral activity of a switch to DOR/ISL compared with continued baseline ART at Week 48. The primary hypothesis is that DOR/ISL is non-inferior to continued baseline ART, as assessed by the percentage of participants with HIV-1 ribonucleic acid (RNA) ≥50 copies/mL at Week 48, with a margin of 4 percentage points used to define non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Is Human Immunodeficiency Virus-1 (HIV-1) positive with plasma HIV-1 Ribonucleic Acid (RNA) <50 copies/mL at screening
* Has been receiving continuous, stable oral 2-drug or 3-drug combination (± PK booster) antiretroviral therapy ART with documented viral suppression (HIV-1 RNA <50 copies/mL) for ≥3 consecutive months prior to providing documented informed consent and has no history of prior virologic treatment failure on any past or current regimen
* Female is not a participant of childbearing potential (POCBP); or if a POCBP uses an acceptable contraceptive method or abstains from penile-vaginal intercourse as their preferred and usual lifestyle; has a negative highly sensitive pregnancy test; and whose medical history, menstrual history, and recent sexual activity has been reviewed by the investigator

Exclusion Criteria:

* Has HIV-2 infection
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has a diagnosis of an active acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within 30 days prior to screening
* Has active hepatitis B virus (HBV) infection
* Has chronic hepatitis C virus (HCV) infection consistent with cirrhosis
* Has a ≤5 years prior history of malignancy
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or strong and moderate cytochrome P450 3A (CYP3A) inducers
* Has taken long-acting HIV therapy at any time
* Is currently participating in or has participated in a clinical study and received (or is receiving) an investigational compound or device from 45 days prior to Day 1 through the study treatment period
* Has a documented or known virologic resistance to Doravine (DOR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2028-07-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (53):
- United States (15):
  - Kaiser Permanente-Infectious Disease ( Site 3014), Los Angeles, California
  - Palmtree Clinical Research ( Site 3032), Palm Springs, California
  - Zuckerberg San Francisco General Hospital and Trauma Center-UCSF ID Clinical Trials Center ( Site 30, San Francisco, California
  - Georgetown University Medical Center ( Site 3006), Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 3009), Ft. Pierce, Florida
  - Orlando Immunology Center ( Site 3004), Orlando, Florida
  - CAN Community Health - Sarasota ( Site 3017), Sarasota, Florida
  - Triple O Research Institute, P.A ( Site 3026), West Palm Beach, Florida
  - Infectious Disease Specialists of Atlanta ( Site 3003), Decatur, Georgia
  - Chatham County Health Department - Chatham CARE Center-Infectious Disease ( Site 3028), Savannah, Georgia
  - ID Care ( Site 3041), Hillsborough, New Jersey
  - Penn Medicine: University of Pennsylvania Health System-Perelman Center for Advanced Medicine ( Site, Philadelphia, Pennsylvania
  - Central Texas Clinical Research ( Site 3015), Austin, Texas
  - The Crofoot Research Center ( Site 3040), Houston, Texas
  - DCOL Center for Clinical Research ( Site 3022), Longview, Texas
- Australia (5):
  - Holdsworth House Medical Practice ( Site 4200), Darlinghurst, New South Wales
  - St Vincent's Hospital-IBAC ( Site 4203), Sydney, New South Wales
  - Holdsworth House Medical Practice - Brisbane ( Site 4201), Brisbane, Queensland
  - Royal Brisbane and Women's Hospital-Infectious Diseases Research ( Site 4204), Brisbane, Queensland
  - Prahran Market Clinic ( Site 4202), Melbourne, Victoria
- Canada (5):
  - Hamilton Health Sciences- Urgent Care Centre-SIS Clinic ( Site 3104), Hamilton, Ontario
  - Maple Leaf Research ( Site 3103), Toronto, Ontario
  - Toronto General Hospital ( Site 3102), Toronto, Ontario
  - Clinique de médecine Urbaine du Quartier Latin ( Site 3101), Montreal, Quebec
  - Clinique Medicale lActuel-Clinical Research ( Site 3100), Montreal, Quebec
- Colombia (3):
  - Ciensalud Ips S A S ( Site 3300), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 3305), Barranquilla, Atlántico
  - Fundacion Valle del Lili- CIC ( Site 3302), Cali, Valle del Cauca Department
- Japan (3):
  - National Hospital Organization Nagoya Medical Center ( Site 4403), Nagoya, Aichi-ken
  - Tokyo Medical University Hospital ( Site 4404), Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 4401), Shinjyuku-ku, Tokyo
- South Africa (9):
  - Josha Research ( Site 3903), Bloemfontein, Free State
  - Perinatal HIV Research Unit (PHRU)-Adult Treatment and Research ( Site 3905), Johannesburg, Gauteng
  - Helen Joseph Hospital ( Site 3910), Johannesburg, Gauteng
  - Ezintsha-Clinical Research Site ( Site 3907), Johannesburg, Gauteng
  - Private Practice Dr. Marleen de Jager ( Site 3900), Pretoria, Gauteng
  - Wentworth Hospital ( Site 3904), Durban, KwaZulu-Natal
  - Family Clinical Research Unit (Fam-Cru)-Adult Infectious Diseases ( Site 3908), Cape Town, Western Cape
  - Desmond Tutu Health Foundation ( Site 3902), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 3901), Paarl, Western Cape
- Switzerland (6):
  - University Hospital Basel-Infectiology ( Site 4002), Basel, Canton of Basel-City
  - Hôpitaux Universitaires de Genève (HUG)-Infectious Disease Department ( Site 4004), Geneva, Canton of Geneva
  - CHUV (centre hospitalier universitaire vaudois) ( Site 4006), Lausanne, Canton of Vaud
  - UniversitätsSpital Zürich ( Site 4000), Zurich, Canton of Zurich
  - Ospedale Regionale di Lugano, Sede Civico-Servizio Malattie Infettive ( Site 4005), Lugano, Canton Ticino
  - Inselspital Bern-Inselspital Infektiologie ( Site 4003), Bern
- United Kingdom (7):
  - Brighton and Sussex University Hospitals NHS Trust ( Site 4104), East Sussex, Brighton And Hove
  - North Manchester General Hospital ( Site 4107), Crumpsall, England
  - Royal London Hospital ( Site 4100), London, England
  - Royal Free Hospital ( Site 4101), London, England
  - Royal Victoria Infirmary ( Site 4105), Newcastle upon Tyne, England
  - King's College Hospital ( Site 4108), London, London, City of
  - Heartlands Hospital ( Site 4102), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Orkin C, Mngqibisa R, Velez JD, Kumar P, Braun DL, Carr A, Bloch M, Walmsley S, Tebas P, Yokomaku Y, Diamond TL, Jackson B, Eves K, Grandhi A, Fuszard M, Klopfer SO, Stamm LM, Fox MC, Kim J. Switch to fixed-dose doravirine (100 mg) and islatravir (0.25 mg) once daily in virologically suppressed adults with HIV-1 on oral antiretroviral therapy: 48-week results of a phase 3, multicentre, randomised, open-label, non-inferiority trial. Lancet. 2026 Feb 7;407(10528):599-610. doi: 10.1016/S0140-6736(25)01945-2. PMID 41654374
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26163&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults living with human immunodeficiency virus-1 (HIV-1) receiving baseline antiretroviral therapy (ART) were enrolled.
Pre-assignment Details: Of the 553 participants randomly assigned in a 2:1 ratio to either Group 1: participants switched from baseline ART to doravirine (DOR)/islatravir (ISL) on Day 1 to Week 144; or Group 2: participants continued baseline ART until Week 48 then switch to DOR/ISL from Week 48 to Week 144, 551 participants received treatment.
Groups:
- Doravirine/Islatravir (DOR/ISL): Participants with Human Immunodeficiency Virus-1 (HIV-1) that have been virologically suppressed for ≥3 consecutive months who were previously treated with continuous baseline antiretroviral therapy (ART) received doravine/islatravir (DOR/ISL), a fixed dose combination (FDC) of 100 mg DOR/0.25 mg ISL orally once daily (qd) for 144 weeks. At Week 144, participants who consent to enter the optional study extension will continue to receive DOR/ISL qd (100 mg/0.25 mg) for an additional 96 weeks or until it is commercially accessible (whichever comes first).
- Baseline ART + DOR/ISL: Participants with HIV-1 that has been virologically suppressed for ≥3 consecutive months who were previously treated with continuous baseline ART received standard of care (SOC) ART for 48 weeks, followed by treatment with DOR/ISL as a FDC of 100 mg DOR/0.25 mg ISL orally qd until Week 144. At Week 144, participants who consent to enter the optional study extension will continue to receive DOR/ISL qd (100 mg/0.25 mg) for an additional 96 weeks or until it is commercially accessible (whichever comes first).
Period: Overall Study
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Started | 368 | 185
Treated | 366 | 185
Completed | 9 | 3
Not Completed | 359 | 182
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Ongoing | 353 | 177
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL | Total
Number analyzed (Participants) | 368 | 185 | 553
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.6) | 49.5 (11.8) | 49.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 67 | 219
  Male | 216 | 118 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 26 | 80
  Not Hispanic or Latino | 310 | 157 | 467
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 18 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 166 | 84 | 250
  White | 143 | 74 | 217
  More than one race | 38 | 16 | 54
  Unknown or Not Reported | 1 | 0 | 1
Baseline Antiretroviral (ART) Stratification at Randomization [Number; unit: Count of Participants] — Participants were stratified into the following baseline ART regimen: (1) Protease inhibitor (PI)-containing regimens (including PI- and integrase strand transferase inhibitor [InSTI]-containing regimens); (2) InSTI-based regimens (non-PI containing regimens); (3) All other non-PI- and non-InSTI containing regimens. Population: All randomized participants who received study intervention.
  Count of Participants
    PI-containing regimens (including PI- and InSTI-containing regimens): number analyzed (Participants) | 366 | 185 | 551
    PI-containing regimens (including PI- and InSTI-containing regimens) | 22 | 8 | 30
    InSTI-based regimens (non-PI containing regimens): number analyzed (Participants) | 366 | 185 | 551
    InSTI-based regimens (non-PI containing regimens) | 233 | 121 | 354
    All other non-PI- and non-InSTI containing regimens: number analyzed (Participants) | 366 | 185 | 551
    All other non-PI- and non-InSTI containing regimens | 111 | 56 | 167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL at Week 48
Description: HIV-1 RNA levels in plasma were measured by polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study intervention and had data for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 366 | 185
Percentage of Participants | 1.4 | 4.9
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Non-Inferiority — Doravirine/Islatravir (DOR/ISL) - Baseline Antiretroviral Therapy (ART). Non-inferiority was concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI was less than 4 percentage points; p < 0.001, Miettinen and Nurminen; The Miettinen and Nurminen method was stratified by corrected baseline ART regimen with Cochran-Mantel-Haenszel (CMH) weights; Estimated difference = -3.58, 95% CI 2-sided [-7.81 to -0.77]

2. Primary Outcome: Percentage of Participants With One or More Adverse Events (AEs) at Week 48
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Day 1 up to Week 48 are reported.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 366 | 185
Percentage of Participants | 79.5 | 83.8
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Other — Difference in percentage versus Baseline Antiretroviral Therapy (ART). Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated difference = -4.3, 95% CI 2-sided [-10.7 to 2.8] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants With an AE Leading to Discontinuation of Study Intervention at Week 48
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE leading to discontinuation of study intervention from Day 1 up to Week 48 are reported.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 366 | 185
Percentage of Participants | 0.5 | 2.2
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated difference = -1.6, 95% CI [-4.9 to 0.2] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 48
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study intervention and had data for analysis excluding participants who had at least one major deviation that may substantially affect the results of the outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 366 | 185
Percentage of Participants | 95.6 | 95.7
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated difference = -0.08, 95% CI [-3.49 to 4.21] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 366 | 185
Percentage of Participants | 95.6 | 91.9
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated difference = 3.75, 95% CI [-0.31 to 8.89] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 96
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 96 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

7. Secondary Outcome: Participants With HIV-1 RNA <200 Copies/mL at Week 144
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 144 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL at Week 96
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 96 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL at Week 144
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 144 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

11. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 144
Description: HIV-1 RNA levels in plasma were measured by a polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 144 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

12. Secondary Outcome: Mean Change of Plasma Cluster of Differentiation 4 (CD4+) T-Cell Count From Baseline Day 1 to Week 48
Description: Plasma CD4+ T-Cell Count was measured in cells/mm^3 for baseline and 48 weeks. Baseline measurements were defined as the Day 1 value of each participant. The mean change of plasma CD4+ T-Cell count from baseline to Week 48 is presented.
Time Frame: Baseline at Day 1 and Week 48
Population: All randomized participants who received at least one dose of study intervention and who have baseline data.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 352 | 178
cells/mm^3 | 5.41 [-12.11 to 22.94] | 18.22 [-11.84 to 48.28]
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; Test type: Other — Difference in mean change from baseline versus Baseline Antiretroviral Therapy (ART); Estimated difference = -15.43, 95% CI [-46.32 to 15.47] — Difference in percentage versus (vs) Baseline ART was based on a cDLA model

13. Secondary Outcome: Mean Change of Plasma CD4+ T-Cell Count From Baseline Week 48 to Week 96
Description: Mean change from baseline at Week 48 in CD4+ T-cell count at Week 96. This outcome measure is applicable to participants who were randomized to switch to DOR/ISL at Week 48.
Time Frame: Baseline at Week 48 and Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

14. Secondary Outcome: Mean Change of Plasma CD4+ T-Cell Count From Baseline Day 48 to Week 144
Description: Mean change from baseline at Week 48 in CD4+ T-cell count at Week 144. This outcome measure is applicable to participants who were randomized to switch to DOR/ISL at Week 48.
Time Frame: Baseline at Week 48 and Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

15. Secondary Outcome: Mean Change of Plasma CD4+ T-Cell Count From Baseline Day 1 to Week 96
Description: Mean change from baseline at Day 1 in CD4+ T-cell count at Week 96. This outcome measure is applicable to those randomized to start DOR/ISL on Day 1.
Time Frame: Baseline at Day 1 and Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

16. Secondary Outcome: Mean Change of Plasma CD4+ T-Cell Count From Baseline Day 1 to Week 144
Description: Mean change from baseline at Day 1 in CD4+ T-cell count at Week 144. This outcome measure is applicable to those randomized to start DOR/ISL on Day 1.
Time Frame: Baseline at Day 1 and Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

17. Secondary Outcome: Percentage of Participants With Treatment-Emergent, Resistance-associated Substitutions at Week 48
Description: Participants with clinically significant confirmed viremia [2 consecutive occurences 4 weeks (+-1 week) apart of HIV-1 RNA >=200 copies/mL at any time during the study] or who discontinue study intervention for another reason with HIV-1 RNA >=200 copies/mL at the time of discontinuation met the criteria for post-baseline resistance testing. Participants with HIV-1 RNA >=400 copies/mL or any participant for whom available genotypic or phenotypic data show evidence of resistance, irrespective of viral load were included in the resistance analysis subset. Plasma samples were collected for genotypic and phenotypic HIV-1 viral drug resistance testing and used to assess resistance-associated substitutions and virus susceptibility to study intervention. The percentage of participants in the resistance analysis subset with treatment-emergent resistance-associated substitutions to the study intervention is presented.
Time Frame: Up to Week 48
Population: Participants with HIV-1 RNA >=400 copies/mL or any participant for whom available genotypic or phenotypic data show evidence of resistance, irrespective of viral load were included in the resistance analysis subset.
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 3 | 0
Percentage of participants | 0 |

18. Secondary Outcome: Mean Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 48
Description: Blood serum samples were taken at baseline and Week 48. The mean change from baseline in fasting Low density lipoprotein cholesterol (LDL-C) at Week 48 is presented for PI-containing regimens (including PI- + InSTI-containing regimens), non-PI- and non-InSTI-containing regimens, and InSTI-containing regimens (non-PI-containing regimens) are presented.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least one dose of study intervention and had baseline data and at least one post-baseline test result in the specified analysis window.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 235 | 129
mg/dL
  PI-containing regimens (including PI- + InSTI-containing regimens): number analyzed (Participants) | 10 | 4
  PI-containing regimens (including PI- + InSTI-containing regimens) | -7.10 [-27.06 to 12.86] | -2.75 [-9.91 to 4.41]
  non-PI- and non-InSTI-containing regimens: number analyzed (Participants) | 69 | 41
  non-PI- and non-InSTI-containing regimens | 5.07 [-0.77 to 10.91] | 0.29 [-5.92 to 6.50]
  InSTI-containing regimens (non-PI-containing regimens): number analyzed (Participants) | 156 | 84
  InSTI-containing regimens (non-PI-containing regimens) | 2.45 [-0.73 to 5.63] | -0.37 [-5.02 to 4.28]
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; PI-containing regimens (including PI- + InSTI-containing regimens); Test type: Superiority — Treatment difference versus baseline ART; p = 0.8340, ANCOVA; Estimated Difference = -2.21, 95% CI 2-sided [-24.91 to 20.49] — The multiplicity adjusted 95% CIs for treatment difference were calculated from ANCOVA models with terms for baseline measurement and treatment
Statistical Analysis 2: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; non-PI- and non-InSTI-containing regimens; Test type: Superiority — Treatment difference versus baseline ART; p = 0.4250, ANCOVA; Estimated Difference = 3.44, 95% CI 2-sided [-5.08 to 11.97] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; InSTI-containing regimens (non-PI-containing regimens); Test type: Superiority — Treatment difference versus baseline ART; p = 0.1618, ANCOVA; Estimated Difference = 3.72, 95% CI [-1.50 to 8.95] — [estimate comment as in outcome 18, analysis 1]

19. Secondary Outcome: Mean Change From Baseline in Fasting Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 48
Description: Blood serum samples were taken at baseline and Week 48. The mean change from baseline in fasting Non-HDL-C at Week 48 is presented for PI-containing regimens (including PI- + InSTI-containing regimens), non-PI- and non-InSTI-containing regimens, and InSTI-containing regimens (non-PI-containing regimens) are presented.
Time Frame: Baseline and Week 48
Population: as for outcome 18
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
Number analyzed (Participants) | 235 | 129
mg/dL
  PI-containing regimens (including PI- + InSTI-containing regimens): number analyzed (Participants) | 10 | 4
  PI-containing regimens (including PI- + InSTI-containing regimens) | -11.80 [-32.04 to 8.44] | -2.75 [-10.90 to 5.40]
  non-PI- and non-InSTI-containing regimens: number analyzed (Participants) | 69 | 41
  non-PI- and non-InSTI-containing regimens | 5.78 [-0.40 to 11.97] | 0.44 [-6.47 to 7.35]
  InSTI-containing regimens (non-PI-containing regimens): number analyzed (Participants) | 156 | 84
  InSTI-containing regimens (non-PI-containing regimens) | 3.60 [0.06 to 7.14] | 3.29 [-5.87 to 12.44]
Statistical Analysis 1: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; PI-containing regimens (including PI- + InSTI-containing regimens); Test type: Superiority — Treatment difference versus baseline ART; Estimated Difference = -7.02, 95% CI 2-sided [-29.80 to 15.77] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; non-PI- and non-InSTI-containing regimens; Test type: Superiority — Treatment difference versus baseline ART; Estimated Difference = 3.99, 95% CI [-5.22 to 13.21] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Doravirine/Islatravir (DOR/ISL) vs Baseline ART + DOR/ISL; InSTI-containing regimens (non-PI-containing regimens); Test type: Superiority — Treatment difference versus baseline ART; Estimated Difference = 1.02, 95% CI 2-sided [-6.83 to 8.87] — [estimate comment as in outcome 18, analysis 1]

20. Secondary Outcome: Participants With One or More AEs at Week 96
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Day 1 up to Week 96 is reported.
Time Frame: Up to Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

21. Secondary Outcome: Participants With One or More AEs at Week 144
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Day 1 up to Week 144 is reported.
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

22. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention at Week 96
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE leading to discontinuation of study intervention from Day 1 up to Week 96 are reported.
Time Frame: Up to Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

23. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention at Week 144
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE leading to discontinuation of study intervention from Day 1 up to Week 144 are reported.
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

24. Secondary Outcome: Percentage of Participants With One or More AEs From Week 48 up to Week 96
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Week 48 up to Week 96 is reported.
Time Frame: Week 48 up to Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

25. Secondary Outcome: Percentage of Participants With One or More AEs From Week 48 up to Week 144
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Week 48 up to Week 144 is presented.
Time Frame: Week 48 up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

26. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention From Week 48 up to Week 96
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE leading to discontinuation of study intervention from Week 48 up to Week 96 are reported.
Time Frame: Week 48 up to Week 96
Reporting Status: Not Posted, anticipated posting 2029-07

27. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention From Week 48 up to Week 144
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE leading to discontinuation of study intervention from Week 48 up to Week 144 are reported.
Time Frame: Week 48 up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-07

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events up to 48 weeks.
Description: All-cause mortality (ACM): all randomized participants; AEs: all randomized participants who received at least one dose of study treatment.
Arm/Group | Doravirine/Islatravir (DOR/ISL) | Baseline ART + DOR/ISL
All-Cause Mortality (participants affected / at risk) | 0/368 | 1/185
Serious Adverse Events (participants affected / at risk) | 23/366 | 9/185
Other Adverse Events (participants affected / at risk) | 123/366 | 73/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine/Islatravir (DOR/ISL) (N=366) | Baseline ART + DOR/ISL (N=185)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine/Islatravir (DOR/ISL) (N=366) | Baseline ART + DOR/ISL (N=185)
Diarrhoea (Gastrointestinal disorders) | 29 (30) | 3 (3)
COVID-19 (Infections and infestations) | 14 (15) | 10 (10)
Nasopharyngitis (Infections and infestations) | 20 (24) | 12 (14)
Upper respiratory tract infection (Infections and infestations) | 38 (45) | 25 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (19) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 10 (10)
Headache (Nervous system disorders) | 19 (21) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT05631093/Prot_SAP_000.pdf